CLINICAL TRIAL: NCT04522011
Title: Comparison of the Efficiency Between Intraoperative and Postoperative Hyperthermic Intraperitoneal Chemotherapy With Docetaxel Combine Oxaliplatin in Patients With Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2019-028
Record Dates: First submitted 2020-08-17; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Stomach Neoplasms; Hyperthermic Intraperitoneal Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: D1/2 radical gastrectomy combines intraoperative hyperthermic intraperitoneal chemotherapy with docetaxel + oxaliplatin
  Interventions: Other: intraoperative or postoperative hyperthermic intraperitoneal chemotherapy
- Group B: D1/2 radical gastrectomy combines postoperative hyperthermic intraperitoneal chemotherapy with docetaxel + oxaliplatin
  Interventions: Other: intraoperative or postoperative hyperthermic intraperitoneal chemotherapy
- Group: without hyperthermic intraperitoneal chemotherapy

INTERVENTIONS:
Other: intraoperative or postoperative hyperthermic intraperitoneal chemotherapy — Intraoperative hyperthermic intraperitoneal chemotherapy：Use docetaxel + oxaliplatin Intraoperately.(Docetaxel 30mg/m2 + oxaliplatin 30mg/m2), perfusion at 43 ℃ for 1 hour
  Groups: Group A; Group B

SUMMARY:
Advanced gastric cancer has always been the focus and difficulty in the treatment of gastric cancer, and postoperative peritoneal recurrence is one of the key factors with poor prognosis. in recent years, hyperthermic intraperitoneal chemotherapy has been used in the treatment of advanced peritoneal metastases and achieved remarkable results. Existing studies have shown that postoperative hyperthermic intraperitoneal chemotherapy plays a certain role in reducing postoperative peritoneal recurrence of advanced gastric cancer. Our previous studies have shown that hyperthermic intraperitoneal chemotherapy adopted docetaxel combine oxaliplatin can also reduce the peritoneal recurrence of advanced gastric cancer. At present, there is a lack of comparison of the safety and efficacy of intraoperative and postoperative hyperthermic intraperitoneal chemotherapy. In this study, patients with advanced gastric cancer were selected by preoperative imaging, endoscopic ultrasonography and other examinations. The patients were randomly divided into group A: D1-2 radical gastrectomy plus hyperthermic intraperitoneal chemotherapy of docetaxel + oxaliplatin. Group B: D1-2 radical gastrectomy + postoperative hyperthermic intraperitoneal chemotherapy of docetaxel + oxaliplatin and group C: D1-2 radical radical gastrectomy .The three groups both proceed postoperative conventional adjuvant chemotherapy（SOX/XELOX）.The incidence of postoperative anastomotic leakage and other complications were collected, and the safety differences among the three groups were compared. The three-year overall survival (OS), disease-free survival (PFS), and disease-related mortality were evaluated and the long-term effects among the three groups were compared.

DETAILED DESCRIPTION:
Background Advanced gastric cancer has always been the focus and difficulty in the treatment of gastric cancer. at present, gastric cancer with clinical stage of T3 / T4a / N + and without distant metastasis is defined as advanced gastric cancer. The conventional treatment is radical surgery plus postoperative or preoperative adjuvant chemotherapy. The overall median survival time is 10-12 months. After surgery-based comprehensive treatment, the 5-year survival rate of advanced gastric cancer is about 30%, and about 30-40% of recurrence is peritoneal recurrence or local recurrence. Postoperative peritoneal recurrence is one of the key factors for poor prognosis of advanced gastric cancer.

Previous peritoneal recurrence and metastasis was defined as the end stage of the disease. Since 1980s, Spratt et al found that chemotherapy combined with hyperthermia can improve the treat efficacy of peritoneal metastases. In the past 20 years, with the progress of accurate temperature control technology, hyperthermic intraperitoneal chemotherapy (HIPEC) has been gradually applied to various advanced peritoneal metastases. HIPEC refers to the accurate constant temperature, circulatory perfusion, filling the abdominal cavity and maintaining for a certain period of time to prevent and treat peritoneal implant metastasis. HIPEC contains three new concepts of precise temperature control, precise positioning and precise removal: (1) accurate temperature control: the accuracy of temperature measurement is less than ±0.1C, the accuracy of temperature control is less than ±0.5C, and the accuracy of flow rate control is less than ±5%. (2) accurate positioning: "x" abdominal cavity cross-placed perfusion tube to the subdiaphragm and pelvic floor to fill the whole abdominal cavity, leaving no treatment blind area, giving full play to the best effect of HIPEC. (3) accurate clearance: volume removal of free cancer cells, subclinical lesions and microcancerous nodules. Intraperitoneal hyperthermic perfusion chemotherapy has been used in the treatment of advanced peritoneal metastases such as gastric cancer, colorectal cancer and ovarian cancer, and achieved remarkable results. The overall prognosis of patients with peritoneal metastases has been greatly improved without increasing adverse reactions.

Research status Previous peritoneal recurrence and metastasis was defined as the end stage of the disease. Since 1980s, Spratt et al found that chemotherapy combined with hyperthermia can improve the treat efficacy of peritoneal metastases. In the past 20 years, with the progress of accurate temperature control technology, hyperthermic intraperitoneal chemotherapy (HIPEC) has been gradually applied to various advanced peritoneal metastases. HIPEC refers to the accurate constant temperature, circulatory perfusion, filling the abdominal cavity and maintaining for a certain period of time to prevent and treat peritoneal implant metastasis. HIPEC contains three new concepts of precise temperature control, precise positioning and precise removal: (1) accurate temperature control: the accuracy of temperature measurement is less than ±0.1C, the accuracy of temperature control is less than ±0.5C, and the accuracy of flow rate control is less than ±5%. (2) accurate positioning: "x" abdominal cavity cross-placed perfusion tube to the subdiaphragm and pelvic floor to fill the whole abdominal cavity, leaving no treatment blind area, giving full play to the best effect of HIPEC. (3) accurate clearance: volume removal of free cancer cells, subclinical lesions and microcancerous nodules. Intraperitoneal hyperthermic perfusion chemotherapy has been used in the treatment of advanced peritoneal metastases such as gastric cancer, colorectal cancer and ovarian cancer, and achieved remarkable results. The overall prognosis of patients with peritoneal metastases has been greatly improved without increasing adverse reactions.

A French analysis of 1125 patients over the past 25 years shows that tumor cell reduction surgery (CRS) combined with hyperthermic intraperitoneal chemotherapy(HIPEC) may benefit patients' survival regardless of the origin of peritoneal metastatic cancer. Foreign GASTRICHIP studies have shown that radical resection of advanced gastric cancer D1-2 gastric cancer plus postoperative hyperthermic intraperitoneal chemotherapy can reduce postoperative peritoneal recurrence of advanced gastric cancer to a certain extent. At present, the HIPEC study of advanced gastric cancer in China is mainly based on the mode of surgery combined with postoperative HIPEC treatment, including the ongoing NCT02381847 study led by Professor Guan Wenxian of Nanjing Gulou Hospital and the NCT03604614 study led by Professor Wang Wei of Guangdong Hospital of traditional Chinese Medicine. both of them are aimed at the safety and efficacy of postoperativehyperthermic intraperitoneal chemotherapy for advanced gastric cancer. At present, there is no clinical study on hyperthermic intraperitoneal chemotherapy at home and abroad.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with gastric adenocarcinoma diagnosed pathologically from 18 to 65 years old.
* 2.Transthoracic and abdominal contrast-enhanced CT and endoscopic ultrasonography were diagnosed as cT3 / T4 N (+).
* 3.There are no obvious surgical taboos in cardiopulmonary function and blood coagulation.
* 4.Ability to provide informed consent

Exclusion Criteria:

* 1.Physical strength score ZPS > = 2.
* 2.Distant metastasis
* 3.Pregnant or lactating.
* 4.Have serious chronic diseases (hypertension, diabetes, etc.).
* 5.Allergic to chemotherapeutic drugs.
* 6.Poor compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who was diagnosed with gastric adenocarcinoma by pathology in the first affiliated Hospital of Jiaotong University since November 2019.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival（0S） | 1 month
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive. In a clinical trial, measuring the overall survival is one way to see how well a new treatment works. Also called OS.
Progression-free survival | 1 month
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. In a clinical trial, measuring the PFS is one way to see how well a new treatment works. Also called progression-free survival.
The incidence of postoperative complications | through study completion, an average of 1 month
  The incidence of medical problems that occurs after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kun Sun, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Kun Zhu, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu J, Huang C, Sun Y, Su X, Cao H, Hu J, Wang K, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Hu Y, Liu H, Zheng C, Li P, Xie J, Liu F, Li Z, Zhao G, Yang K, Liu C, Li H, Chen P, Ji J, Li G; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Effect of Laparoscopic vs Open Distal Gastrectomy on 3-Year Disease-Free Survival in Patients With Locally Advanced Gastric Cancer: The CLASS-01 Randomized Clinical Trial. JAMA. 2019 May 28;321(20):1983-1992. doi: 10.1001/jama.2019.5359. PMID 31135850
- [Background] Yonemura Y, Elnemr A, Endou Y, Hirano M, Mizumoto A, Takao N, Ichinose M, Miura M, Li Y. Multidisciplinary therapy for treatment of patients with peritoneal carcinomatosis from gastric cancer. World J Gastrointest Oncol. 2010 Feb 15;2(2):85-97. doi: 10.4251/wjgo.v2.i2.85. PMID 21160926
- [Background] Glehen O, Passot G, Villeneuve L, Vaudoyer D, Bin-Dorel S, Boschetti G, Piaton E, Garofalo A. GASTRICHIP: D2 resection and hyperthermic intraperitoneal chemotherapy in locally advanced gastric carcinoma: a randomized and multicenter phase III study. BMC Cancer. 2014 Mar 14;14:183. doi: 10.1186/1471-2407-14-183. PMID 24628950
- [Background] Yonemura Y, Elnemr A, Endou Y, Ishibashi H, Mizumoto A, Miura M, Li Y. Effects of neoadjuvant intraperitoneal/systemic chemotherapy (bidirectional chemotherapy) for the treatment of patients with peritoneal metastasis from gastric cancer. Int J Surg Oncol. 2012;2012:148420. doi: 10.1155/2012/148420. Epub 2012 Jul 31. PMID 22900159
- [Background] Roviello F, Caruso S, Marrelli D, Pedrazzani C, Neri A, De Stefano A, Pinto E. Treatment of peritoneal carcinomatosis with cytoreductive surgery and hyperthermic intraperitoneal chemotherapy: state of the art and future developments. Surg Oncol. 2011 Mar;20(1):e38-54. doi: 10.1016/j.suronc.2010.09.002. Epub 2010 Dec 15. PMID 20888755
- [Background] Helm JH, Miura JT, Glenn JA, Marcus RK, Larrieux G, Jayakrishnan TT, Donahue AE, Gamblin TC, Turaga KK, Johnston FM. Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy for malignant peritoneal mesothelioma: a systematic review and meta-analysis. Ann Surg Oncol. 2015 May;22(5):1686-93. doi: 10.1245/s10434-014-3978-x. Epub 2014 Aug 15. PMID 25124472
- [Background] Bonnot PE, Piessen G, Kepenekian V, Decullier E, Pocard M, Meunier B, Bereder JM, Abboud K, Marchal F, Quenet F, Goere D, Msika S, Arvieux C, Pirro N, Wernert R, Rat P, Gagniere J, Lefevre JH, Courvoisier T, Kianmanesh R, Vaudoyer D, Rivoire M, Meeus P, Passot G, Glehen O; FREGAT and BIG-RENAPE Networks. Cytoreductive Surgery With or Without Hyperthermic Intraperitoneal Chemotherapy for Gastric Cancer With Peritoneal Metastases (CYTO-CHIP study): A Propensity Score Analysis. J Clin Oncol. 2019 Aug 10;37(23):2028-2040. doi: 10.1200/JCO.18.01688. Epub 2019 May 14. PMID 31084544